CLINICAL TRIAL: NCT00138398
Title: T-cell Responses Predict Influenza Risk in Older Adults
Brief Title: T-cell Response-Flu Risk in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 05-0056
Record Dates: First submitted 2005-08-26; First posted 2005-08-30 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2013-02

CONDITIONS: Influenza
Keywords: Influenza, T cell, vaccine, Congestive heart failure
MeSH Terms: conditions — Influenza, Human; Heart Failure

INTERVENTIONS:
Biological: Commercial TriValent Split Influenza Virus

SUMMARY:
The purpose of this study is to determine how the immune system changes with aging and makes influenza a more serious illness in older people. Influenza vaccination not only can protect people from getting the flu but also can lessen the severity of the illness. This is particularly true for people with congestive heart failure (CHF). This research may provide information that could eventually lead to a new laboratory test that will predict how effective vaccination is for preventing influenza illness in older people. Volunteer participants in this study will include the following groups: 1) healthy young adults 20 - 40 years old; 2) older adults, 60 years and older, without a history of CHF; 3) older adults, 60 years and older, with a history of CHF. All study participants will be vaccinated with the current preparation of inactivated influenza vaccine. A small amount of blood will be drawn before each vaccine and at 4, 10, and 16-20 weeks afterward.

DETAILED DESCRIPTION:
This study will increase the understanding of how age, congestive heart failure (CHF) or a prior hospitalization for an influenza-related acute coronary event affect the immune response to influenza vaccination. By elucidating the defects in the immune response to influenza vaccination that are associated with the subsequent influenza illness, these methods can be used to screen subsets of older adults to establish the risk profile related to influenza in that population, to target these defects for future vaccine development and to use these methods as surrogates of protection to screen potential vaccines prior to conducting large scale clinical trials to establish clinical efficacy. The primary objective is to show that granzyme B (Grz B) levels in influenza virus-stimulated peripheral blood mononuclear cell cultures are lower in older adults who receive inactivated influenza vaccine (IIV) and subsequently develop influenza illness compared to those who do not. Secondary objectives are to: (1) establish a cut-off value for Grz B as a marker of increased risk for influenza illness; (2) show that interferon-gamma (IFN-gamma) levels are lower and interleukin-10 (IL-10) levels are higher in influenza virus-stimulated peripheral blood mononuclear cell cultures from vaccinated older adults who subsequently develop influenza illness compared to those who do not; (3) determine the effect of macrophage migration inhibitory facator (MIF) on T-cell responses to influenza vaccination; (4) determine the association between CHF and ischemic heart disease (IHD) including acute coronary syndromes and the immune response to influenza vaccination; (5) determine the effect of functional status measured by the Six-Minute Walk Test (SMWT) on immune responsiveness to influenza vaccination; (6) determine the effect of medications with anti-inflammatory effects including angiotensin converting enzyme inhibitors (ACEI) and cholesterol-lowering drugs (statins) on immune responsiveness to influenza vaccination; (7) evaluate the effect of the age-related decline in the expression of the costimulatory molecule, CD28, on cytotoxic T-lymphocytes, on the Grz B response to influenza vaccination; (8) study the potential role of activation-induced cell death (AICD) on the T helper type 1 (Th1: IFN-gamma) versus T helper type 2 (Th2: IL-10) response to influenza vaccination; (9) determine in vitro whether or not co-stimulatory molecules such as 4-1BB ligand or CD70 can be used to augment the cytokine, Grz B or CTL responses to influenza vaccines in older adults; (10) determine in vitro whether or not heat shock proteins (HSP) can be used to augment the cytokine and/or Grz B response to influenza vaccination in older adults; (11) determine in vitro whether or not heat shock proteins (HSP) can be used to augment the cytokine and/or Grz B response to influenza vaccination in older adults who develop influenza illness in spite of influenza vaccination; and (12) determine in vitro whether or not heat shock proteins (HSP) increase the frequency, Grz B content or proportion of influenza virus-specific CTL expressing CD28 in vaccinated in older adults. The study group will consist of 150 adults, age 60 years and older, characterized according to age, presence of CHF or IHD, or (to be identified in the prior influenza season) an admission with an acute coronary syndrome or exacerbation of CHF. All subjects will be vaccinated in the fall of each year with the current preparation of trivalent, split-virus influenza vaccine. Serum antibody titers, serum cytokine levels, ex vivo levels of IFN-gamma and IL-10, and ex vivo and in vitro levels of Grz B in influenza-stimulated peripheral blood mononuclear cell at pre-vaccination and post-vaccination (4, 10 and 16-20 weeks) time points will be compared in subjects who do and do not get influenza illness. The peak as well as the duration of response to vaccination for each of the immunologic measures will be determined.

ELIGIBILITY:
Inclusion Criteria:

* Willing to be vaccinated with the current influenza vaccine.
* Healthy young adults are 20-40 years and have no underlying chronic diseases.
* 'Healthy' older adult participants are age 60 and older who may have underlying chronic diseases but no diagnosis of CHF, advanced kidney disease or diabetes requiring insulin.
* High-risk older adults with cardiovascular disease are age 60 years and older and have a diagnosis of CHF, or IHD including ACS in the previous winter season.

Exclusion Criteria:

* Allergic reactions to eggs or preservatives such as those contained in contact lens solutions.
* A previous significant reaction to vaccination or if they refuse to receive influenza vaccination.
* Known immunosuppressive disorders or medications (including oral prednisone in doses >10 mg daily) or have not received influenza vaccination in the past.
* Subjects who report respiratory illness within the two-week period prior to vaccination. Subjects reporting respiratory symptoms at the first study visit are re-scheduled to a time when they have not had a respiratory illness (at least two symptoms of cough, runny nose, malaise and fever) within the two-week period prior to vaccination.
* Cardiovascular diseases due to intravenous drug abuse, myocarditis or congenital abnormalities
* Any condition that in the opinion of the investigator would interfere with the interpretation or the evaluation of the vaccine

Ages: 20 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 850
Dates: Start 2005-10-25

CONTACTS AND LOCATIONS:
Locations (1):
- University of Connecticut Health Center, Farmington, Connecticut, United States